CLINICAL TRIAL: NCT01799304
Title: Is it Possible to Improve Static and Dynamic Postural Stability in Cerebral Palsy Children by Modulating Attention?
Brief Title: Static and Dynamic Postural Stability in Cerebral Palsy Children
Acronym: Dual-Task
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DCIC - 13 01
Record Dates: First submitted 2013-02-14; First posted 2013-02-26 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: CP (Cerebral Palsy); Diplegia; Hemiplegia; Postural; Defect
Keywords: Locomotion; cerebral palsy; Postural; Defect
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- no distractor control group (Experimental): postural control and locomotion of CP children without attentional distractor and without additional cognitive task (control condition)
  Interventions: Procedure: no distractor control group
- visual and sound attentional distractors (Experimental): postural control and locomotion of CP children with visual and sound attentional distractors (video film).
  Interventions: Procedure: visual and sound attentional distractors
- sound attentional distractor alone (Experimental): postural control and locomotion of CP children with sound attentional distractor alone (sound track of the video film).
  Interventions: Procedure: sound attentional distractor alone
- additional cognitive task (Experimental): postural control and locomotion of CP children with an additional cognitive task (adapted Stroop task with animals)
  Interventions: Procedure: additional cognitive task

INTERVENTIONS:
Procedure: no distractor control group — This control condition will aim at analyzing posture and locomotion in CP children with the intent to focus attention on their equilibrium, only, without any other interference.
  Arms: no distractor control group
Procedure: visual and sound attentional distractors — The distractors will be used to orient subjects' attention toward another simple and motivating task in order to avoid focalisation on postural control and locomotion and to favour a more automatic control.
  Arms: visual and sound attentional distractors
Procedure: sound attentional distractor alone — In addition to the previous condition, the goal of the present condition is to isolate the effects of a sound distractor, since it is known that CP children frequently exhibit visual deficits which may affect their postural and locomotion difficulties.
  Arms: sound attentional distractor alone
Procedure: additional cognitive task — The additional cognitive task aimed to increase the attentional load and to analyse its impact on children's capacity to process two tasks simultaneously (the cognitive and postural or locomotor tasks)
  Arms: additional cognitive task

SUMMARY:
Cerebral palsy (CP) concerns 2 children out of 1000 in the general population (SCPE 2002). It is the main cause of postural and motor deficits in children.

During the past 20 years, the postural deficits exhibited by these children have been attributed to various factors :

1. neuromuscular functions
2. sensory integration
3. muscular-squeletic functions.

The common point of all these studies is the existence of immature motor patterns, probably related to an inability to implement more elaborated and adapted motor patterns with respect the task to perform.

CP children do not develop the characteristics of the plant grad locomotion. They exhibit a uniform muscular activation with a high level of co-activation. Locomotion is generally characterized by an increase of stretching reflexes at short latencies and by a low level of activation associated to a low modulation of gastrocnemius muscles..

These data also suggest that it is the control of the temporal rather than the spatial parameters of the head which are mainly altered in CP children.

Even though static postural control and locomotion are considered as automatic processes, this control requires, however, a significant amount of attentional resources.

Within this context, the amount of attentional resources which need to be solicited can provide information on two complementary dimensions. On one hand, on the level of automaticity of postural control and/or locomotion when subjects' attention is oriented toward another task. On the other hand, on the cognitive cost of postural control and/or locomotion, depending on children age, that is, as a function of their level of maturation and of the nature and importance of their sensory-motor deficits. When the amount of required attentional resources is reduced, postural control and/or locomotion is considered as automatic processes with a low cognitive cost.

The dual task paradigm in which subjects have to simultaneously process a cognitive (e.g. Stroop task) and a postural or motor task (e.g., standing upright on a force platform) is generally used to investigate these questions.

How an appropriate allocation of attention is performed as a function of the cognitive and postural/motor tasks is important in the developmental process of posture and locomotion. It seems to be even more crucial in CP children and more generally in pathology.

The main goal of the present project is to investigate the contribution of attentional processes in postural control and locomotion of CP children as compared to control healthy children.

DETAILED DESCRIPTION:
Within this scientific and clinical context, we hypothesize:

* That CP children will be less stable than healthy children (in control situation) and that the attentional cost for controlling static posture will be higher.
* On the basis of Olivier et al.'s work (2008) showing in adults and children aged 4 to 11 that postural control is better when attention is oriented toward a video film (i.e., decrease of the attentional demand allocated to the control of static posture), we predict that CP children will be more stable in dual task situation with visual or sound distractors than when focusing attention on postural control alone.
* We also predict that an additional cognitive task (adapted Stroop task), by increasing the attentional demand, will induce a deficit of postural control confirming Reilly et al.'s results (2008b).

On the same basis, we will also investigate the attentional cost of locomotion.

Exploratory study of dynamic equilibrium during locomotion in the same conditions.

Investigation of posture in the following conditions:

1. without attentional distractors and without additional cognitive task (control condition)
2. with attentional visual and sound distractors (video film)
3. with sound attentional distractor alone (sound track of the video film)
4. with an additional cognitive task (Stroop task adapted for children).

Considering the goals of this research project, no serious undesirable event is expected to occur. However, falls may occur accidentally while rising or descending from the force platform, during static posture, or during locomotion. Consequently, in addition to the experimenter, a physiotherapist or someone of the medical staff will be present during all experimental recordings.

The environment will be also organized to the secure the experimental room by excluding all potentials dangerous or non necessary objects. Whenever necessary, the potentials falls will be reported and declared to the health authorities.

ELIGIBILITY:
Inclusion Criteria:

* CP children with postural and/or motor deficits due to early cerebral deficits (from conception to 2 years of age according to G. Tardieu) non hereditary and non evolutionary.
* Aged 7 to 12 years because before 7 years of age the range and speed of postural control exhibit a great variability and after 12, our eligibility criteria are not standardized
* presenting a clinical CP diplegia or hemiplegia (cf. EMGF),
* able to stand upright without assistance for at least (real recording time of 30 sec during the experiment) on a force platform (L 50 cm x l 50 cm x h 4,4 cm) and to walk straight ahead on a walking track (518 cm long x 90 cm wide and 0,5 cm thin) without assistance,
* without severe visual or hearing deficit (>0,3 for the worse eye without correction or hearing loss <70db for the worse ear without correction) as indicated in the personal medical report
* without hyperactivity trouble (Conners' questionnaires non significant <70), without major attentional deficits (images matching test), without denomination troubles (ELOLA test), able to perform dual tasks (Tea-ch test).

Exclusion Criteria:

* parents' or children' informed consent rejected,
* Participation to another biomedical experiment during this study,
* Children unable to control upright posture without assistance for at least 45 sec on a force platform (L 50 cm x l 50 cm x h 4.4 cm) or unable to walk without assistance
* Absence of social security coverage.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The main goal of the present project is to investigate the contribution of attentional processes in postural control and locomotion of CP children as compared to control healthy children. | First day of inclusion T0
  Mean velocity of center of foot pressure displacements (mm/sec) in static posture under the different experimental conditions

SECONDARY OUTCOMES:
Without attentional distractor and without additional cognitive task (control condition) | First day of inclusion T0
  This control condition will aim at analyzing posture and locomotion in CP children with the intent to focus attention on their equilibrium, only, without any other interference.
  Outcome measurement : Mean velocity of center of foot pressure displacements (mm/sec)
With visual and sound attentional distractors (video film). | First day of inclusion T0
  The distractors will be used to orient subjects' attention toward another simple and motivating task in order to avoid focalisation on postural control and locomotion and to favour a more automatic control.
  Outcome measurement : Mean velocity of center of foot pressure displacements (mm/sec)
With sound attentional distractor alone (sound track of the video film). | First day of inclusion T0
  In addition to the previous condition, the goal of the present condition is to isolate the effects of a sound distractor, since it is known that CP children frequently exhibit visual deficits which may affect their postural and locomotion difficulties.
  Outcome measurement : Mean velocity of center of foot pressure displacements (mm/sec)
With an additional cognitive task (adapted Stroop task with animals). | First day of inclusion T0
  The additional cognitive task aimed to increase the attentional load and to analyse its impact on children's capacity to process two tasks simultaneously (the cognitive and postural or locomotor tasks) Outcome measurement : Mean velocity of center of foot pressure displacements (mm/sec)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine COMMARE, MD, Principal Investigator — Unité de MPR Pédiatrique, CHU GRENOBLE; Vincent NOUGIER, Pr, Principal Investigator — Laboratoire TIMC-IMAG, Faculté de Médecine; Dominic PÉRENNOU, Pr, Principal Investigator — Clinique MPR- Institut de Rééducation- Hôpital sud, CHU Grenoble; Isabelle OLIVIER, Pr, Principal Investigator — Laboratoire TIMC-IMAG, Faculté de Médecine; BARBIERI GUILLAUME, Study Chair — Laboratoire TIMC-IMAG, Faculté de Médecine; FARIGOULE VINCENT, MD, Principal Investigator — University Hospital, Grenoble; PRADO CHLOE, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble, Grenoble, France

REFERENCES:
- [Background] Agostini, M., Metz-Lutz , M.N., Van Hout, A., Chavance, M., Deloche, G., Pavao- Martins & Dellatolas. 1998. Batterie d'évaluation du langage oral de l'enfant aphasique - ELOLA. Revue de Neuropsychologie, 8, 319-367
- [Background] Albaret, JM., Benesteau, J., & Marquet-Doleac J. 1999. AI Test d'appariement d'images. Éditions ECPA
- [Background] Berger W, Altenmueller E, Dietz V. Normal and impaired development of children's gait. Hum Neurobiol. 1984;3(3):163-70. PMID 6480437
- [Background] Berger W. Characteristics of locomotor control in children with cerebral palsy. Neurosci Biobehav Rev. 1998 Jul;22(4):579-82. doi: 10.1016/s0149-7634(97)00047-x. PMID 9595572
- [Background] Blanchard Y, Carey S, Coffey J, Cohen A, Harris T, Michlik S, Pellecchia GL. The influence of concurrent cognitive tasks on postural sway in children. Pediatr Phys Ther. 2005 Fall;17(3):189-93. doi: 10.1097/01.pep.0000176578.57147.5d. PMID 16357673
- [Background] Brogren E, Hadders-Algra M, Forssberg H. Postural control in sitting children with cerebral palsy. Neurosci Biobehav Rev. 1998 Jul;22(4):591-6. doi: 10.1016/s0149-7634(97)00049-3. PMID 9595574
- [Background] Burtner PA, Qualls C, Woollacott MH. Muscle activation characteristics of stance balance control in children with spastic cerebral palsy. Gait Posture. 1998 Dec 1;8(3):163-174. doi: 10.1016/s0966-6362(98)00032-0. PMID 10200406
- [Background] Cherng RJ, Su FC, Chen JJ, Kuan TS. Performance of static standing balance in children with spastic diplegic cerebral palsy under altered sensory environments. Am J Phys Med Rehabil. 1999 Jul-Aug;78(4):336-43. doi: 10.1097/00002060-199907000-00008. PMID 10418839
- [Background] Christ SE, White DA, Brunstrom JE, Abrams RA. Inhibitory control following perinatal brain injury. Neuropsychology. 2003 Jan;17(1):171-8. PMID 12597086
- [Background] Crenna P, Inverno M, Frigo C, Palmieri R, Fedrizzi E. Pathophysiological profile of gait in children with cerebral palsy. In: Forssberg H, hirschfeld H, editors. Movement disorders in children. Karger: Medicine and Sport Sciences. Basel; 1992. p. 186-98.
- [Background] Crenna P, Inverno M. Objective detection of pathophysiological factors contributing to gait disturbance. In motor development in children, E. Fedrizzi, G. Avanzini and P. Crenna. John Libbey (Eds) London;1994. p. 103-18.
- [Background] Crenna P. Spasticity and 'spastic' gait in children with cerebral palsy. Neurosci Biobehav Rev. 1998 Jul;22(4):571-8. doi: 10.1016/s0149-7634(97)00046-8. PMID 9595571
- [Background] Heinen F, Desloovere K, Schroeder AS, Berweck S, Borggraefe I, van Campenhout A, Andersen GL, Aydin R, Becher JG, Bernert G, Caballero IM, Carr L, Valayer EC, Desiato MT, Fairhurst C, Filipetti P, Hassink RI, Hustedt U, Jozwiak M, Kocer SI, Kolanowski E, Krageloh-Mann I, Kutlay S, Maenpaa H, Mall V, McArthur P, Morel E, Papavassiliou A, Pascual-Pascual I, Pedersen SA, Plasschaert FS, van der Ploeg I, Remy-Neris O, Renders A, Di Rosa G, Steinlin M, Tedroff K, Valls JV, Viehweger E, Molenaers G. The updated European Consensus 2009 on the use of Botulinum toxin for children with cerebral palsy. Eur J Paediatr Neurol. 2010 Jan;14(1):45-66. doi: 10.1016/j.ejpn.2009.09.005. Epub 2009 Nov 14. PMID 19914110
- [Background] Holt KG, Ratcliffe R, Jeng SF. Head stability in walking in children with cerebral palsy and in children and adults without neurological impairment. Phys Ther. 1999 Dec;79(12):1153-62. PMID 10630284
- [Background] Lajoie Y, Teasdale N, Bard C, Fleury M. Attentional demands for static and dynamic equilibrium. Exp Brain Res. 1993;97(1):139-44. doi: 10.1007/BF00228824. PMID 8131825
- [Background] Laufer Y, Ashkenazi T, Josman N. The effects of a concurrent cognitive task on the postural control of young children with and without developmental coordination disorder. Gait Posture. 2008 Feb;27(2):347-51. doi: 10.1016/j.gaitpost.2007.04.013. Epub 2007 May 29. PMID 17532635
- [Background] Leonard C. Neural and behavioral changes associated with perinatal damage. In: H.Forssberg and H. Hirschfeld Eds. Movement Disorders in Children. Karger: Medicine and Sport Science Basel; 1992. p. 50-6.
- [Background] Lowes LP, Westcott SL, Palisano RJ, Effgen SK, Orlin MN. Muscle force and range of motion as predictors of standing balance in children with cerebral palsy. Phys Occup Ther Pediatr. 2004;24(1-2):57-77. doi: 10.1300/j006v24n01_03. PMID 15268998
- [Background] Mainly T., Robertson IH, Anderson V., & Mimmo-Smith I. 2004. Test d'évaluation de l'attention chez l'enfant. Éditions ECPA
- [Background] Molin I, Alricsson M. Physical activity and health among adolescents with cerebral palsy in Sweden. Int J Adolesc Med Health. 2009 Oct-Dec;21(4):623-33. doi: 10.1515/ijamh.2009.21.4.623. PMID 20306774
- [Background] Nashner LM, Shumway-Cook A, Marin O. Stance posture control in select groups of children with cerebral palsy: deficits in sensory organization and muscular coordination. Exp Brain Res. 1983;49(3):393-409. doi: 10.1007/BF00238781. PMID 6641837
- [Background] Okoshi Y, Itoh M, Takashima S. Characteristic neuropathology and plasticity in periventricular leukomalacia. Pediatr Neurol. 2001 Sep;25(3):221-6. doi: 10.1016/s0887-8994(01)00309-5. PMID 11587877
- [Background] Olivier I, Cuisinier R, Vaugoyeau M, Nougier V, Assaiante C. Dual-task study of cognitive and postural interference in 7-year-olds and adults. Neuroreport. 2007 May 28;18(8):817-21. doi: 10.1097/WNR.0b013e3280e129e1. PMID 17471073
- [Background] Olivier I, Cuisinier R, Vaugoyeau M, Nougier V, Assaiante C. Age-related differences in cognitive and postural dual-task performance. Gait Posture. 2010 Oct;32(4):494-9. doi: 10.1016/j.gaitpost.2010.07.008. Epub 2010 Aug 9. PMID 20692161
- [Background] Olivier I, Palluel E, Nougier V. Effects of attentional focus on postural sway in children and adults. Exp Brain Res. 2008 Feb;185(2):341-5. doi: 10.1007/s00221-008-1271-6. Epub 2008 Jan 24. PMID 18214449
- [Background] Palluel E, Nougier V, Olivier I. Postural control and attentional demand during adolescence. Brain Res. 2010 Oct 28;1358:151-9. doi: 10.1016/j.brainres.2010.08.051. Epub 2010 Aug 22. PMID 20735993
- [Background] Platt MJ, Cans C, Johnson A, Surman G, Topp M, Torrioli MG, Krageloh-Mann I. Trends in cerebral palsy among infants of very low birthweight (<1500 g) or born prematurely (<32 weeks) in 16 European centres: a database study. Lancet. 2007 Jan 6;369(9555):43-50. doi: 10.1016/S0140-6736(07)60030-0. PMID 17208641
- [Background] Reilly DS, van Donkelaar P, Saavedra S, Woollacott MH. Interaction between the development of postural control and the executive function of attention. J Mot Behav. 2008 Mar;40(2):90-102. doi: 10.3200/JMBR.40.2.90-102. PMID 18400676
- [Background] Reilly DS, Woollacott MH, van Donkelaar P, Saavedra S. The interaction between executive attention and postural control in dual-task conditions: children with cerebral palsy. Arch Phys Med Rehabil. 2008 May;89(5):834-42. doi: 10.1016/j.apmr.2007.10.023. PMID 18452729
- [Background] Seidman LJ, Valera EM, Makris N, Monuteaux MC, Boriel DL, Kelkar K, Kennedy DN, Caviness VS, Bush G, Aleardi M, Faraone SV, Biederman J. Dorsolateral prefrontal and anterior cingulate cortex volumetric abnormalities in adults with attention-deficit/hyperactivity disorder identified by magnetic resonance imaging. Biol Psychiatry. 2006 Nov 15;60(10):1071-80. doi: 10.1016/j.biopsych.2006.04.031. Epub 2006 Jul 28. PMID 16876137
- [Background] Prevalence and characteristics of children with cerebral palsy in Europe. Dev Med Child Neurol. 2002 Sep;44(9):633-40. PMID 12227618
- [Background] Woollacott MH, Burtner P. Neural and musculoskeletal contributions to the development of stance balance control in typical children and in children with cerebral palsy. Acta Paediatr Suppl. 1996 Oct;416:58-62. doi: 10.1111/j.1651-2227.1996.tb14279.x. PMID 8997450
- [Background] Woollacott MH, Burtner P, Jensen J, Jasiewicz J, Roncesvalles N, Sveistrup H. Development of postural responses during standing in healthy children and children with spastic diplegia. Neurosci Biobehav Rev. 1998 Jul;22(4):583-9. doi: 10.1016/s0149-7634(97)00048-1. PMID 9595573
- [Background] Woollacott MH, Crenna P. Postural control in standing and walking in children with cerebral palsy. Chapter. In: Hadders-Algra M, Brogren Carlberg E, editors. Posture: a key issue in developmental disorders. London: Mac Keith Press; 2008.